CLINICAL TRIAL: NCT06663033
Title: COVID-19 Specific Risk Factor for Anastomotic Leak After Colorectal Cancer Surgery. a Retrospective Study
Brief Title: Anastomotic Leak in Covid-19
Status: Completed | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Tamer.A.A.M.Habeeb, professour of general and laparoscopic surgery, Zagazig University
Other Study IDs: anastomotic leak
Record Dates: First submitted 2024-10-27; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Anastomosis, Leaking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | US Export: No

INTERVENTIONS:
Procedure: colorectal surgery — surgery for colorectal cancer

SUMMARY:
evaluate the incidence of anastomotic leak after colorectal surgery

ELIGIBILITY:
Inclusion Criteria:

* colorectal cancer

Exclusion Criteria:

* stage 4

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with colorectal cancer
Sampling Method: Probability Sample
Enrollment: 390 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
anastomotic leak | 30 days
  incidence of anastomotic leak

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Zagazig University, Zagazig, Sharqia Province, Egypt